CLINICAL TRIAL: NCT04695288
Title: Relationship Between Kinesiophobia, Quality of Life, and Cognitive Functions in Fibromyalgia Syndrome
Brief Title: Kinesiophobia, Quality of Life, and Cognitive Functions in Fibromyalgia Syndrome
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Şeniz Akçay, Study Director, Bozyaka Training and Research Hospital
Other Study IDs: 01/12/2020-297
Record Dates: First submitted 2021-01-02; First posted 2021-01-05 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Fibromyalgia; Kinesiophobia; Cognitive Dysfunction
Keywords: Fibromyalgia; Kinesiophobia; Cognition; Quality of life
MeSH Terms: conditions — Fibromyalgia; Kinesiophobia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia Syndrome: 100 participants with a diagnosis of Fibromyalgia Syndrome according to the 2016 revised American College of Rheumatology diagnostic criteria.
- Control subjects: 60 healthy participants do not meet the exclusion criteria of the study.

SUMMARY:
Although one of the most evidence-based treatment protocols is based on exercise strategies in patients with Fibromyalgia Syndrome, fear and avoidance of physical activity; named 'Kinesiophobia' may hinder the patients from the exercises. Cognitive dysfunctions are seen frequently in Fibromyalgia Syndrome. The aim of this study, to assess the relationship between kinesiophobia and cognitive functions, disease severity, quality of life, physical activity level, pain intensity, and anxiety/depression level in Fibromyalgia patients. Additionally, the investigators aimed to compare the kinesiophobia level and cognitive functions between patients with Fibromyalgia Syndrome and control subjects.

DETAILED DESCRIPTION:
Cognitive dysfunction, including learning difficulties, memory, attention, and executive dysfunctions are frequent in fibromyalgia syndrome. Kinesiophobia is defined as fear and avoidance of physical activities, and it can lead to increased disability in patients with chronic pain. Although there is a relationship between cognitive functions and physical performance in Fibromyalgia Syndrome, the relationship between kinesiophobia, fibrofog, and quality of life are required to be investigated.

The aims of this study are:

1. To compare the kinesiophobia and cognitive functions in Fibromyalgia Syndrome with healthy volunteers
2. To examine the relationship between the severity of kinesiophobia, cognitive functions, disease activity, quality of life, physical activity level, depression and anxiety severity in Fibromyalgia Syndrome.

The hypothesis is, the patients diagnosed with Fibromyalgia Syndrome have higher kinesiophobia severity and worse cognitive functions, and also that kinesiophobia severity is associated with cognitive dysfunction, disease severity, physical activity level, and psychiatric symptoms in patients with Fibromyalgia Syndrome.

ELIGIBILITY:
Inclusion Criteria:

-Fibromyalgia Syndrome

Exclusion Criteria:

* Education year < 5
* Inflammatory rheumatic disease
* Malignancy
* Psychiatric disease
* Alcohol/substance addiction
* Central nervous system disease
* History of head trauma
* Chronic pain conditions other than Fibromyalgia Syndrome

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Fibromyalgia Syndrome is more common in women than in men. For this reason, we predicted that there might be inequality in the distribution of male/female in the participant group included.
  Physical activity level and psychiatric scales may differ between genders.
Study Population: Fibromyalgia Syndrome participants and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
TAMPA Kinesiophobia Scale | 1 year
  The TAMPA Kinesiophobia Scale consists of 17 questions. Each question is scored between 1-4. The maximum score is 68, with high scores indicating an increased severity of kinesiophobia. A score of more than 37 indicates high severity of kinesiophobia.
Montreal Cognitive Assessment Test | 1 year
  This test evaluates eight separate cognitive functions: Attention, working memory, short-term memory, delayed memory, visuospatial abilities, executive functioning, language, and orientation to time and place. Scores of 21 and above are considered normal, with the highest test score being 30.

SECONDARY OUTCOMES:
Visual Analogue scale | 1 year
  The patient is asked to mark her severity of pain on a horizontal 10-cm line with number 0 on one end representing "no" and number 10 on the other end indicating "very severe pain". Higher scores indicate higher levels of pain intensity.
Fibromyalgia Impact Questionnaire | 1 year
  It aims to evaluate the arthritis symptoms and functional status of patients with fibromyalgia syndrome through 21 questions that inquire about physical functions, work-related situations, depression, anxiety, waking up tired, pain, stiffness, and fatigue. Higher scores indicate greater impact of fibromyalgia on functioning. Final score should range from 0 to 80.
Short Form-36 | 1 year
  Short Form-36 (SF-36) is a widely used and validated scale for evaluating the quality of life. It is not specific to any disease group. It consists of thirty six items. It consists of 8 subscales related to physical health (physical function, physical role, pain, general health) and mental health (energy, social function, emotional role difficulty, mental health) factors. Each sub-scale chart is evaluated between 0 and 100 points. Higher scores indicate good health.
International Physical Activity Questionnaire-Short Form | 1 year
  Physical activity levels in the last 7 (seven) days will be evaluated with the International Physical Activity Questionnaire-Short form. This short form consists of seven questions and provides information about the durations of physical activities, walking and sitting within the last seven days in the metabolic equivalent (MET)-min/week unit.
Hospital Anxiety/ Depression Questionnaire | 1 year
  Hospital Anxiety/ Depression Questionnaire determines the risk in terms of anxiety and depression in the patient and to measure its level and severity. It is used to diagnose anxiety and depression in a short time and determine the risk group for patients with physical diseases and those who apply to primary health care. Seven (odd numbers) of 14 questions measure anxiety and seven (even numbers) measure depression. Answers are scored in a four-point Likert scale between 0 and 3. The lowest score that patients can get from both subscales is 0, the highest score is 21.

CONTACTS AND LOCATIONS:
Overall Officials: Elcin Ergez, MD, Principal Investigator — University of Health Sciences Izmir Bozyaka Training and Research Hospital; Seniz Akcay, Assoc Prof, Study Director — University of Health Sciences Izmir Bozyaka Training and Research Hospital; Nesibe Dogan, Specialist, Study Chair — University of Health Sciences Izmir Bozyaka Training and Research Hospital; Dursun Hakan Delibas, Specialist, Study Chair — University of Health Sciences Izmir Bozyaka Training and Research Hospital
Locations (1):
- University of Health Sciences Izmir Bozyaka Training and Research Hospital, Izmir, Karabaglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The clinical study report will be shared at the end of the study.

REFERENCES:
- [Background] Mease P. Fibromyalgia syndrome: review of clinical presentation, pathogenesis, outcome measures, and treatment. J Rheumatol Suppl. 2005 Aug;75:6-21. PMID 16078356
- [Background] Katz RS, Heard AR, Mills M, Leavitt F. The prevalence and clinical impact of reported cognitive difficulties (fibrofog) in patients with rheumatic disease with and without fibromyalgia. J Clin Rheumatol. 2004 Apr;10(2):53-8. doi: 10.1097/01.rhu.0000120895.20623.9f. PMID 17043464
- [Background] Denison E, Asenlof P, Lindberg P. Self-efficacy, fear avoidance, and pain intensity as predictors of disability in subacute and chronic musculoskeletal pain patients in primary health care. Pain. 2004 Oct;111(3):245-252. doi: 10.1016/j.pain.2004.07.001. PMID 15363867
- [Background] KoCyIGIt BF, Akaltun MS. Kinesiophobia Levels in Fibromyalgia Syndrome and the Relationship Between Pain, Disease Activity, Depression. Arch Rheumatol. 2020 Feb 7;35(2):214-219. doi: 10.46497/ArchRheumatol.2020.7432. eCollection 2020 Jun. PMID 32851370
- [Background] Turk DC, Robinson JP, Burwinkle T. Prevalence of fear of pain and activity in patients with fibromyalgia syndrome. J Pain. 2004 Nov;5(9):483-90. doi: 10.1016/j.jpain.2004.08.002. PMID 15556826
- [Background] Russek L, Gardner S, Maguire K, Stevens C, Brown EZ, Jayawardana V, Mondal S. A cross-sectional survey assessing sources of movement-related fear among people with fibromyalgia syndrome. Clin Rheumatol. 2015 Jun;34(6):1109-19. doi: 10.1007/s10067-014-2494-5. Epub 2014 Jan 31. PMID 24481649